CLINICAL TRIAL: NCT06981689
Title: Association of Breast Reconstruction Method With Long-term Risk of Psychiatric Disorders: A Target Trial Emulation
Brief Title: Association of Breast Reconstruction Method With Long-term Risk of Psychiatric Disorders
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Danbee Kang, Associate Professor, Samsung Medical Center
Other Study IDs: AR vs. IBR
Record Dates: First submitted 2025-04-23; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
Keywords: autologous reconstruction; implant-based reconstruction; psychiatric disorders
MeSH Terms: conditions — Breast Neoplasms; Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- autologous reconstruction: autologous reconstruction following mastectomy
- implant-based reconstruction: implant-based reconstruction following mastectomy

SUMMARY:
Female breast cancer patients who underwent total mastectomy followed by breast reconstruction

DETAILED DESCRIPTION:
Female breast cancer patients who underwent total mastectomy followed by breast reconstruction

ELIGIBILITY:
Inclusion Criteria:

* The study included newly diagnosed female breast cancer patients who underwent total mastectomy

Exclusion Criteria:

* individuals who underwent reconstruction prior to mastectomy
* those diagnosed with psychiatric disorders within one year prior to surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biologically female
Study Population: The study included newly diagnosed female breast cancer patients who underwent total mastectomy followed by breast reconstruction classified into two types using ICD-10 procedure codes: autologous tissue reconstructions were coded from N7140 to N7147 and implant-based reconstructions were coded from N7148 to N7151 Exclusions applied to males, individuals who underwent reconstruction prior to mastectomy, and those diagnosed with psychiatric disorders within one year prior to surgery
Sampling Method: Non-Probability Sample
Enrollment: 24930 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Psychiatric disorders | 1 year, 5 year and 9 year since surgery
  The primary endpoint was clinically diagnosed psychiatric disorder, defined as the first occurrence of a diagnosis made by a physician for any of the following major psychiatric conditions: anxiety disorders (F40, F41), bipolar disorder (F30, F31, F34.0), depressive disorders (F32, F33), sleep disorders (G47.0, F51.0), obsessive-compulsive disorder (F42), posttraumatic stress disorder (F43.1), and substance use disorders (F10-F19).

IPD SHARING:
Plan to Share IPD: No